CLINICAL TRIAL: NCT00496990
Title: Treating the Partners of Drug Using Pregnant Women: Stage II
Acronym: HOPE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Hendree E. Jones, Adjunct Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DA013496 (NIH); R01DA013496 (NIH); DPMCDA
Record Dates: First submitted 2007-07-05; First posted 2007-07-06 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Drug Addiction
Keywords: male; female; couple; cocaine; opiate; methadone; detoxification; pregnancy
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (Active Comparator): Participants in this group receive the opportunity to attend a support group
  Interventions: Behavioral: control
- Enhanced care (Experimental): Participants in this arm receive the opportunity to have detoxification or methadone treatment as well as receive vouchers contingent upon drug free urine samples and individualized counseling
  Interventions: Behavioral: Enhanced care

INTERVENTIONS:
Behavioral: Enhanced care — this group received counseling, contingency management and methadone or detoxification
  Arms: Enhanced care
Behavioral: control — this group receives the opportunity to participate in a support group
  Arms: control

SUMMARY:
This is a two group randomized design that will compare a novel therapy package (i.e., Research supported treatment intervention, Contingency-based voucher incentives for the male partner's drug abstinence, Specialized MI couples counseling) to standard care for helping drug using partners of drug dependent pregnant women obtain and maintain drug abstinence. Participants will be followed for 22 weeks and have scheduled twice weekly urine sample collection and all participants will have follow-up interviews post-study entry.

ELIGIBILITY:
Inclusion Criteria:

* are 18 years of age or older on admission;
* Pregnant as determined by sonogram results
* have a current sexual partner who they have seen recently at least 3 times a week
* male partner has regular alcohol or illicit drug use (at least 4 of 7 days typical use) and is not incarcerated.

Exclusion Criteria:

* woman or partner report current suicidal ideation
* woman or partner meet diagnostic criteria for a current DSM-IV Axis I thought disorder (i.e. schizophrenia)
* woman or partner demonstrate significant cognitive impairment that precludes them from completing the initial assessment battery
* woman has evidence of physical violence or abuse

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 158 (Actual)
Dates: Start 2005-10; Primary Completion 2009-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Partner Objective Substance Use | treatment entry until 28 weeks later

SECONDARY OUTCOMES:
Woman's drug use will be measured with urine toxicology | treatment entry until 28 weeks later

CONTACTS AND LOCATIONS:
Overall Officials: Hendree Jones, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Center for Addiction and Pregnancy Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Lund IO, Kirtadze I, Otiashvili D, O'Grady KE, Jones HE. Female partners of opioid-injecting men in the Republic of Georgia: an initial characterization. Subst Abuse Treat Prev Policy. 2012 Nov 16;7:46. doi: 10.1186/1747-597X-7-46. PMID 23157895
- [Derived] Kirtadze I, Otiashvili D, O'Grady KE, Jones HE. Behavioral treatment + naltrexone reduces drug use and legal problems in the Republic of Georgia. Am J Drug Alcohol Abuse. 2012 Mar;38(2):171-5. doi: 10.3109/00952990.2011.643996. Epub 2012 Jan 5. PMID 22221277
- [Derived] Jones HE, Tuten M, O'Grady KE. Treating the partners of opioid-dependent pregnant patients: feasibility and efficacy. Am J Drug Alcohol Abuse. 2011 May;37(3):170-8. doi: 10.3109/00952990.2011.563336. Epub 2011 Mar 17. PMID 21410418